CLINICAL TRIAL: NCT04793672
Title: A Multi-center Observational Clinical Study Observing the Differences of Tongue Images Between Patients With Malignant Tumors and Healthy People
Brief Title: Establishment of Tongue Image Database and Machine Learning Model for Malignant Tumors Diagnosis
Status: Completed | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other); Zhejiang Hospital of TCM (Unknown); Wenzhou Medical University (Other); Fujian Cancer Hospital (Other Government); RenJi Hospital (Other); Tongde Hospital of Zhejiang (Unknown); Kecheng District People's Hospital (Unknown); Yueyang Central Hospital (Other); Shandong Cancer Hospital and Institute (Other); Shanxi Province Cancer Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Harbin Cancer Hospital (Unknown); Yuhang District People's Hospital (Unknown); Hainan Cancer Hospital (Other); Zigong Fourth People's Hospital (Unknown); Henan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Professor; Chief physician, Zhejiang Cancer Hospital
Other Study IDs: IRB-2019-56
Record Dates: First submitted 2021-03-05; First posted 2021-03-11 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Malignant Tumor
Keywords: Malignant tumor; Tongue Image
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with malignant tumors and healthy people: Tongue images, coating on the tongue and clinical data of patients with malignant tumors and healthy people will be collected.
  Interventions: Other: Tongue images, coating on the tongue and clinical data of patients with malignant tumors and healthy people will be collected.

INTERVENTIONS:
Other: Tongue images, coating on the tongue and clinical data of patients with malignant tumors and healthy people will be collected. — Tongue images, coating on the tongue and clinical data of patients with malignant tumors and healthy people will be collected.

SUMMARY:
The tongue images of malignant tumors and corresponding healthy people will be collected to establish the tongue image database. Deep learning will be carried out by computer and artificial intelligence to construct the early screening, diagnosis, prognosis and prognosis model of various malignant tumors based on tongue image for the diagnosis and treatment of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* 18≤age≤80
* Histologically or cytologically confirmed malignant tumor
* No prior chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor treatment for malignant tumor
* Subject volunteers to join the study, Signs informed consent, has good compliance and can cooperate with follow-up

Exclusion Criteria:

* Two or more kinds of malignant tumors at the same time
* Malignant tumor that has been treated by chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor therapy
* Subjects who had other factors that might force them to terminate the research ahead of time, such as the development of other severe disease (including mental disease) that required combined treatment, seriously abnormal laboratory examination value, and family or social factors that might affect the subject safety or experimental data collection, as judged by the researchers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically confirmed malignant tumor，and no prior chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor treatment for malignant tumor.
Sampling Method: Non-Probability Sample
Enrollment: 4100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The differences of tongue images between patients with malignant tumors and healthy people. | 1 year
Overall Survival (OS) | 3 years

SECONDARY OUTCOMES:
Disease free survival（DFS） | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Cheng, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (2):
- China (2):
  - Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No